CLINICAL TRIAL: NCT07089719
Title: Bevacizumab in Post-acute Sequelae of COVID-19 : Efficacy and Safety (Pilot Study)
Acronym: BASECOVID
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government); ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP241020; RECHMIE-23-0004 (Other Grant/Funding Number: Ministry of health, France); 2024-520308-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-21; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Dyspnea Caused by 2019-nCoV
Keywords: dyspnea caused by 2019-nCov; Covid-19; bevacizumab
MeSH Terms: conditions — COVID-19 | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab (Experimental): Participants will receive Bevacizumab at a dose of 10mg/kg via intravenous infusion. They will receive a total of 5 injections, administered every two weeks.
  Interventions: Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: Bevacizumab Injection — Participants will receive Bevacizumab at a dose of 10mg/kg via intravenous infusion. They will receive a total of 5 injections, administered every two weeks.

SUMMARY:
The aim of this research is to evaluate an innovative treatment, Bevacizumab, in patients suffering from respiratory complications related to COVID-19. These complications, particularly difficulty breathing (dyspnea) and impaired lung function, are common in some individuals after infection. The study seeks to determine whether Bevacizumab can improve breathing capacity by acting on vascular mechanisms that may be responsible for these issues. A total of 21 patients with these persistent symptoms will be included in the study, with close medical monitoring to assess both the effectiveness of the treatment and its safety.

This research aims to assess the effectiveness and safety of Bevacizumab, a medication known for its anti-angiogenic properties (which prevent the formation of new blood vessels), in patients experiencing persistent respiratory problems after COVID-19 infection. In other words, this research is based on the idea that inhibiting blood vessel formation with Bevacizumab may improve clinical outcomes in patients with severe forms of COVID-19 by reducing vascular complications associated with the infection.

To answer this research question, 21 individuals with persistent respiratory symptoms (significant dyspnea) and reduced lung diffusing capacity (DLCO less than 75% of the predicted value) at least three months after their initial COVID-19 infection will be included. The study is being conducted at Hôpital Européen Georges Pompidou, in Paris.

The total expected duration of the research is 31 months, and each patient's participation will last 7 months, which includes 2 months of treatment (five Bevacizumab injections) followed by five additional months of medical follow-up.

In this research project, we will be evaluating Bevacizumab, an experimental drug in the context of Long COVID. Bevacizumab is a monoclonal antibody used to inhibit angiogenesis (the abnormal formation of new blood vessels). While commonly used in oncology, in this study, its use aims to improve lung function in patients suffering from persistent respiratory complications after COVID-19 infection.

Bevacizumab will be administered as an intravenous infusion. The infusion lasts between 30 and 90 minutes. The dosage is 10 mg/kg every two weeks, for a total of five infusions over a two-month period. Additional follow-up visits will be conducted one month and five months after the end of treatment. Monitoring will include clinical examinations, laboratory tests, and lung function assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years, under 90 years
* Social security affiliation
* Good understanding of the French language
* Written informed consent
* DOcumented COVID-19 infection (PCR or CT-scan) more than 3 months before inclusion
* Long COVID suspicion with dyspnea (mMRC > 2 at inclusion)
* DLCO < 75% of predicted value less than 3 months old on the day of screening or to be obtained before Day 1 older than 3 months

Exclusion Criteria:

* Acute COVID-19 infection
* Lung scintigraphy and thoracic CT angiography evaluation to rule out pulmonary embolism less than 3 months old on the day of screening or to be obtained before Day 1 if older than 3 months to exclude Sequelae of pulmonary embolism or lung emphysema in the setting of COPD
* Women of childbearing potential
* Myocardial infarction or stroke less than 3 months before screening
* Uncontrolled hypertension (> 140/90 at inclusion in the study)
* Proteinuria/creatinuria ratio > 1 g/mmol at baseline DFG < 30 ml/min
* History of malignant hypertension
* Previous osteonecrosis
* History of Aneurysm and artery dissections
* Active cancer
* Known hypersensitivity to bevacizumab or any ingredient in its formulation, including non-medicinal ingredients, or a component of the container
* Hypersensitivity to Chinese Hamster Ovary (CHO) cell product or other recombinant human or humanized antibodies
* History of radiotherapy
* History of bisphosphonates treatment
* Surgery in 28 days before inclusion
* Participation in another interventional study or being in the exclusion period at the end of a previous study
* Patient unable or unwilling to comply with the follow up schedule (at the investigator's discretion)
* Pregnant or breastfeeding women
* Vulnerable populations (patient under gardianship, curatorship, deprived of liberty)
* Patient on AME (State medical aid)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with 10% increase of impaired DLCO | 3 months after the introduction of bevacizumab.
  Assess efficacy of bevacizumab injection in long COVID patients with impaired DLCO (<75% of predicted value). The positive criteria will be a 10% increase in DLCO at three months after the introduction of bevacizumab.

SECONDARY OUTCOMES:
Proportion of patients with recovery of clinical symptoms | 1, 2, 3 and 7 months after the initiation of Bevacizumab.
  Modification of clinical evaluation and in particular the clinical symptom of dyspnea and fatigue or other related clinical parameters of long-COVID patients (mMRC Scale, Borg Scale, STOP-BANG Questionnaire, WHODAS 2.0, Epworth Sleepiness Scale, which assess fatigue severity in long-COVID patients).
Proportion of patients with recovery of psychological, cognitive, and autonomic functions | 3 and 7 months after the initiation of Bevacizumab treatment.
  Evaluation of psychological, cognitive, and autonomic functions. In particular, additional assessments will be conducted to evaluate psychological, cognitive, and autonomic functions with the Nijmegen Questionnaire, the Hospital Anxiety and Depression Scale, the Montreal Cognitive Assessment, the self-reported Ricci-Gagnon Physical Activity Questionnaire, the Somatic Symptom Disorder Scale-12 (SSD-12) and the Survey of Autonomic Symptoms.
Proportion of patients with improvement of other parameter than DLCO explored by Pulmonary Function Test | 1, 2, 3 and 7-months after the initiation of Bevacizumab treatment.
  Modification of other respiratory function markers: forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), FEV1/FVC ratio, total lung capacity (TLC), residual volume (RV), and 6-minutes walking distance test between baseline and follow-up.
Modification of DLCO | 1 and 2 months after the initiation of Bevacizumab treatment.
  Difference of DLCO between baseline and follow-up.
Circulating angiogenic biomarkers levels | 1, 2, 3 and 7 months after the initiation of Bevacizumab treatment.
  Difference of circulating angiogenic biomarkers levels between baseline and follow-up.
Number of side effects related to bevacizumab | From bevacizumab treatment initiation to the end of the follow-up at 7 months.
  Safety of bevacizumab in long-COVID patients regarding treatment side effects.
Number of patients with hospitalization or medical consultation | From bevacizumab treatment initiation to the end of the follow-up at 7 months.
  Safety of bevacizumab in long-COVID patients regarding hospitalization or medical consultation.

CONTACTS AND LOCATIONS:
Overall Officials: David Smadja, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - HEGP, clinical investigation center, Paris
  - HEGP, department of Physiology, Paris

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific involvement of the PI team. Collaboration will be fostered.
  Teams wishing obtain IPD must meet the sponsor and IP team to present scientifics (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).

REFERENCES:
- [Background] Philippe A, Gunther S, Rancic J, Cavagna P, Renaud B, Gendron N, Mousseaux E, Hua-Huy T, Reverdito G, Planquette B, Sanchez O, Gaussem P, Salmon D, Diehl JL, Smadja DM. VEGF-A plasma levels are associated with impaired DLCO and radiological sequelae in long COVID patients. Angiogenesis. 2024 Feb;27(1):51-66. doi: 10.1007/s10456-023-09890-9. Epub 2023 Aug 1. PMID 37526809